CLINICAL TRIAL: NCT07227792
Title: Tongue-out Radiation Therapy (TORT) for the Mitigation of Radiotherapy-related Toxicities in Patients With Head and Neck Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yvonne Mowery (Other)
Collaborators: Radiological Society of North America (Other)
Responsible Party: Sponsor-Investigator, Yvonne Mowery, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 25-085
Record Dates: First submitted 2025-11-10; First posted 2025-11-13 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Carcinoma
Keywords: Tongue-out radiation therapy (TORT); human papillomavirus (HPV)-related oropharyngeal cancer; Intensity modulated radiotherapy (IMRT); volumetric modulated arc therapy (VMAT)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Tongue-out radiation therapy (TORT) (Experimental): A treatment positioning technique for patients with head and neck tumors at particular subsites (e.g., oropharynx, larynx, hypopharynx). Protruding the tongue, i.e. "tongue-out" position, during pre-treatment simulation and subsequent treatment induces anatomical changes that facilitate decreased radiation dose to the oral tongue and PCM. All patients will be treated with IMRT. All IMRT techniques, including static field IMRT, helical IMRT (Tomotherapy), and VMAT are allowed.
  Interventions: Radiation: Tongue-out radiation therapy (TORT)

INTERVENTIONS:
Radiation: Tongue-out radiation therapy (TORT) — The high-risk PTV will contain the primary tumor and any lymph nodes confirmed or suspected to harbor metastatic disease based on imaging findings, pathology reports, and/or clinical exam. Dose to the high-risk PTV must be 70.0 Gy at 2.0 Gy per fraction.
  The intermediate-risk PTV will contain areas considered to contain potential microscopic disease in close proximity to the primary tumor (GTV + 10 mm with adjustments per above based on anatomic boundaries or air) and the entire cervical lymph node level(s) corresponding to any lymph nodes confirmed or suspected to harbor metastatic disease. Dose to intermediate-risk PTV must be 63 Gy at 1.8 Gy per fraction.
  The low-risk PTV will contain any cervical lymph node levels felt to be potentially harbor microscopic disease but with negative imaging and/or clinical findings. The exact cervical lymph node levels included in the low-risk PTV should be based on Tables 3-5. Dose to the low-risk PTV must be 56 Gy at 1.6 Gy per fraction.

SUMMARY:
Our institution recently began incorporating a novel "tongue-out" radiation therapy (TORT) technique for patients with head and neck tumors at particular subsites (oropharynx, larynx, hypopharynx). Protruding the tongue, i.e. "tongue-out" position, induces anatomical changes that facilitate decreased radiation dose to the oral tongue and PCM. The long-term goal is to determine whether TORT results in reduced severity and faster recovery from acute treatment-related toxicities (particularly mucositis, dysphagia, and dysgeusia) and improved long-term swallowing function and taste compared to traditional "tongue-in" RT for patients with HNC.

DETAILED DESCRIPTION:
Despite good disease control and organ preservation outcomes after radiotherapy (RT) for head and neck cancers (HNC), particularly human papillomavirus (HPV)-related oropharyngeal cancer, treatment-related toxicities remain a challenging survivorship problem. Impaired calorie intake due to common RT-associated toxicities such as mucositis, dysphagia (difficulty swallowing), and dysgeusia (taste loss) can lead to treatment breaks that reduce treatment efficacy and prolong recovery, some of which persist long-term and negatively impact quality of life (QOL). Radiation doses to the pharyngeal constrictor muscles (PCM) and oral tongue correlate with incidence and severity of dysphagia and dysgeusia. Doses to the pharyngeal and oral tongue mucosa are associated with incidence and severity of mucositis. "Tongue-out" radiation therapy (TORT) is a treatment positioning technique for patients with head and neck tumors at particular subsites (e.g., oropharynx, larynx, hypopharynx). Protruding the tongue, i.e. "tongue-out" position, during pre-treatment simulation and subsequent treatment induces anatomical changes that facilitate decreased radiation dose to the oral tongue and PCM. TORT for oropharyngeal, laryngeal, and hypopharyngeal cancers may result in significantly lower radiation dose to the PCM and oral tongue compared to "tongue-in" RT, and that this reduced dose to organs at risk (OARs) will yield clinically meaningful improvements in severity and duration of dysphagia, dysgeusia, and mucositis.

ELIGIBILITY:
Inclusion Criteria:

1. Must have histologically or cytologically confirmed squamous cell carcinoma of the oropharynx, larynx, or hypopharynx (cT0-4, N0-3, M0-1).
2. Patients with metastatic disease will be included if the following criteria are met:

   * Definitive RT dose is planned for the primary site
   * The number of metastatic lesions is ≤5
   * All metastatic lesions are confined to a single organ (e.g., lung)
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2
4. Female subjects of childbearing potential must not be pregnant or breastfeeding at screening.

   * Female subjects are considered to be of childbearing potential unless one of the following criteria is met:

     o Permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. Note: Documentation may include review of medical records, medical examination, or medical history interview by study site staff.
   * Female subjects of childbearing potential must utilize an appropriate method of birth control such as hormonal methods (oral, injectable, implant, skin patch, vaginal ring), intrauterine devices, barrier methods (consistent use of male/female condoms, diaphragms, cervical caps), surgical methods (vasectomy, tubal ligation), or true abstinence.
5. Must be able to comfortably protrude tongue in the treatment position for at least 1 minute.
6. Must have the ability to understand and the willingness to sign a written informed consent document.
7. Must be willing to comply with all study procedures.
8. Must be able to complete patient-reported outcome (PRO) questionnaires in English.

Exclusion Criteria:

1. Patients with T1-T2 N0 glottic cancer (i.e., planned to undergo RT to the larynx only)
2. Posterior pharyngeal wall primary tumor
3. Widely metastatic disease
4. Surgical resection of the primary tumor
5. Induction chemotherapy or immunotherapy prior to planned radiotherapy
6. Prior head and neck radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-11-23 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Eating Assessment Tool 10 (EAT-10) | At Baseline
  Mean difference in Eating Assessment Tool 10 (EAT-10) total scores between patients enrolled on this prospective study and matched retrospective controls. EAT-10 screens for dysphagia and aspiration risk. Total score ranges 0 - 40. Patients rate each question on a scale of 0 (no problem) to 4 (severe problem) regarding, weight loss, inability to go out for meals, increased swallowing effort, pain while swallowing, reduced pleasure while eating, bolus sensation, coughing, and stress when swallowing. Score of 15 or more means patient is at risk for aspiration. Follow up with a full dysphagia assessment and introduce safe swallowing strategies and a modified diet, as needed. Score of 16 or less means patient may not be at risk for aspiration and follow up with a full dysphagia assessment only if symptomatic.
Eating Assessment Tool 10 (EAT-10) | At 6 weeks post-treatment
  Mean difference in Eating Assessment Tool 10 (EAT-10) total scores between patients enrolled on this prospective study and matched retrospective controls. EAT-10 screens for dysphagia and aspiration risk. Total score ranges 0 - 40. Patients rate each question on a scale of 0 (no problem) to 4 (severe problem) regarding, weight loss, inability to go out for meals, increased swallowing effort, pain while swallowing, reduced pleasure while eating, bolus sensation, coughing, and stress when swallowing. Score of 15 or more means patient is at risk for aspiration. Follow up with a full dysphagia assessment and introduce safe swallowing strategies and a modified diet, as needed. Score of 16 or less means patient may not be at risk for aspiration and follow up with a full dysphagia assessment only if symptomatic.

SECONDARY OUTCOMES:
Eating Assessment Tool 10 (EAT-10) | At 58 weeks post treatment
  Mean difference between EAT-10 scores post-RT for the prospective TORT patients and matched historical controls at this timepoint. EAT-10 screens for dysphagia and aspiration risk. Total score ranges 0 - 40. Patients rate each question on a scale of 0 (no problem) to 4 (severe problem) regarding, weight loss, inability to go out for meals, increased swallowing effort, pain while swallowing, reduced pleasure while eating, bolus sensation, coughing, and stress when swallowing. Score of 15 or more means patient is at risk for aspiration. Follow up with a full dysphagia assessment and introduce safe swallowing strategies and a modified diet, as needed. Score of 16 or less means patient may not be at risk for aspiration and follow up with a full dysphagia assessment only if symptomatic.
Change in Eating Assessment Tool 10 (EAT-10) Scores | At Baseline and 6 weeks post-treatment
  Mean change in EAT-10 scores post-RT for the prospective TORT patients and matched historical controls. EAT-10 screens for dysphagia and aspiration risk. Total score ranges 0 - 40. Patients rate each question on a scale of 0 (no problem) to 4 (severe problem) regarding, weight loss, inability to go out for meals, increased swallowing effort, pain while swallowing, reduced pleasure while eating, bolus sensation, coughing, and stress when swallowing. Score of 15 or more means patient is at risk for aspiration. Follow up with a full dysphagia assessment and introduce safe swallowing strategies and a modified diet, as needed. Score of 16 or less means patient may not be at risk for aspiration and follow up with a full dysphagia assessment only if symptomatic.
Change in Eating Assessment Tool 10 (EAT-10) Scores | At Baseline and 58 weeks post treatment
  Mean change in EAT-10 scores between for the prospective TORT patients and matched historical controls. EAT-10 screens for dysphagia and aspiration risk. Total score ranges 0 - 40. Patients rate each question on a scale of 0 (no problem) to 4 (severe problem) regarding, weight loss, inability to go out for meals, increased swallowing effort, pain while swallowing, reduced pleasure while eating, bolus sensation, coughing, and stress when swallowing. Score of 15 or more means patient is at risk for aspiration. Follow up with a full dysphagia assessment and introduce safe swallowing strategies and a modified diet, as needed. Score of 16 or less means patient may not be at risk for aspiration and follow up with a full dysphagia assessment only if symptomatic.
University of Washington Quality of Life Questionnaire (UW-QOL) | At 6 weeks post-treatment
  Mean difference between UW-QOL swallowing scores post-RT for the prospective TORT patients and matched historical controls at this timepoint. Self-administered UW-QOL measures health and quality of life over prior 7 days. 12 domain-specific questions include a patient's evaluation of the following: pain, appearance, activity, recreation, swallowing, chewing, speech, shoulder, taste, saliva, mood, and anxiety. The UW-QOL domains are based upon discrete ordinal responses. Scoring is scaled to so that a score of 0 represents the worst possible response, and a score of 100 represents the best possible response. Scoring is scaled in equal stages from 0 to 100 to reflect the number of possible responses.
Change in QoL per University of Washington Quality of Life Questionnaire (UW-QOL) | At Baseline and 6 weeks post-treatment
  Mean change in UW-QOL swallowing scores for the prospective TORT patients and matched historical controls. Self-administered UW-QOL measures health and quality of life over prior 7 days. 12 domain-specific questions include a patient's evaluation of the following: pain, appearance, activity, recreation, swallowing, chewing, speech, shoulder, taste, saliva, mood, and anxiety. The UW-QOL domains are based upon discrete ordinal responses. Scoring is scaled to so that a score of 0 represents the worst possible response, and a score of 100 represents the best possible response. Scoring is scaled in equal stages from 0 to 100 to reflect the number of possible responses.
Difference in radiation doses - oral tongue | Up to 38 months
  Mean difference in radiation doses (number of Gy) to the oral tongue as measured in radiation treatment planning software between TORT and non-TORT plans for the same patients.
Difference in radiation doses - pharyngeal | Up to 38 moonths
  Mean difference in radiation doses (number of Gy) to the pharyngeal constrictors muscles as measured in radiation treatment planning software between TORT and non-TORT plans for the same patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Mowery, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No